CLINICAL TRIAL: NCT01521988
Title: Prevention of Atrial Fibrillation by Combined Right Isthmus Ablation and cryoBalloon Pulmonary Vein Isolation in Patients With Typical Atrial Flutter
Brief Title: Cryoballoon Pulmonary Venous Isolation in Patients Referred for Typical Atrial Flutter Ablation
Acronym: PAF CRIOBLAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011/089/HP
Record Dates: First submitted 2011-11-28; First posted 2012-01-31 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Atrial Flutter; Atrial Fibrillation
Keywords: Atrial flutter; Atrial fibrillation; Catheter ablation
MeSH Terms: conditions — Atrial Flutter; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atrial flutter ablation (Active Comparator): RF atrial flutter ablation
  Interventions: Procedure: Atrial flutter ablation
- Atrial flutter ablation and pulmonary vein isolation (Experimental): RF Atrial flutter ablation and pulmonary vein isolation using cryoablation
  Interventions: Procedure: Atrial flutter ablation and pulmonary vein isolation

INTERVENTIONS:
Procedure: Atrial flutter ablation — Radiofrequency ablation of Atrial flutter
  Arms: Atrial flutter ablation
Procedure: Atrial flutter ablation and pulmonary vein isolation — Radiofrequency ablation of atrial flutter and pulmonary vein isolation using cryoablation
  Arms: Atrial flutter ablation and pulmonary vein isolation

SUMMARY:
- Background:

Atrial fibrillation is frequently associated with typical atrial flutter in clinical practice. If the radical treatment of atrial flutter by radiofrequency catheter is achieved in most cases without recurrence, it does not prevent the occurrence of atrial fibrillation that occurs in about 70% of these patients after several years of follow-up. However, the latter arrhythmia is associated with significant morbidity and mortality. The problem of atrial fibrillation occurrence after successful ablation of typical atrial flutter remains physicians primary concern in monitoring these patients.

* Objectives:

The purpose of this study is to demonstrate that the pulmonary veins isolation using balloon cryotherapy technology performed at the time of flutter ablation, significantly reduces the risk of developing atrial fibrillation in the two year period following the procedure.

* Selection Criteria:

Patients referred for ablation of typical atrial flutter with an history of at least one documented episode of atrial fibrillation (atrial flutter remaining the predominant arrhythmia)will be enrolled in the study.

* Study Methods:

This is a prospective, multicenter, randomized, 2-arms study, comparing the rate of atrial fibrillation occurrence over a two years period following either an ablation procedure of typical atrial flutter (Group 1), or a combined procedure of typical atrial flutter ablation and pulmonary veins cryoballoon isolation (Group 2). The enrollment period will be of 18 months.

Randomization will be 1:1 and will be balanced in blocks of varying size. Patients will then be regularly followed up clinically and by long-term ECG recordings.

* Evaluation Criteria:

The primary endpoint will be the recurrence of symptomatic or asymptomatic atrial fibrillation, documented by an ECG or an R-test, occurring between M3 and M24

* Number of patients:

  170 patients will be enrolled in the study
* Number of centers:

Four French and three German centers will participate.

* Perspective:

The demonstration of a clinical benefit in terms of atrial fibrillation risk reduction in the patient group with pulmonary vein isolation, could lead to a modification of atrial arrhythmia treatment indication.

ELIGIBILITY:
* Inclusion Criteria:

  * Patient with a spontaneous flutter or with a flutter recurrence when it was not considered appropriate to use a preventive treatment so far. The flutter may have been paroxysmal or may still be present.
  * Patient with at least one documented episode of typical flutter defined as follows: negative F waves in the inferior territory, positive in V1 and negative in V6 lead, F wave pattern with characteristic "saw tooth" appearance and finally a heart rate comprised between 240 and 320 beats per minute.
  * Patient with effective anticoagulant therapy for at least 3 weeks.
  * Patient with at least one episode of AF (lasting more than 1 minute) documented on an ECG or a 24 hour Holter recording
  * Patient who signed an informed consent.
  * Patient with age ≥ 18 yo and ≤ 75 yo
* Exclusion Criteria:

  * Patients with the following characteristics will be excluded:

    * Contraindication to right-heart catheterization
    * Contraindication to an anticoagulant treatment
    * Patient for which AF is predominant (more recordings of AF than Flutter)
    * Persistent AF at the time of inclusion visit
    * History of mitral valve surgery
    * Known disorders of blood clotting
    * Cardiothyreosis
  * Life expectancy < 24 months
  * Less than 18 years old and pregnant ladies. As before any ablation, a pregnancy test will be done the day before or the day of the procedure
  * Patient less than 18 years old
  * Patient under guardianship
  * Patient deprived of their liberty by a court decision

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Recurrence of symptomatic or asymptomatic AF as documented on an ECG or a long term Holter | an average of 24 months following the ablation procedure
  Main endpoint will be the recurrence of symptomatic or asymptomatic atrial fibrillation as documented by an ECG or a R-test. Sustained AF episodes of more than a minute will be classified depending if they are symptomatic or not.

SECONDARY OUTCOMES:
Recurrence rate of typical atrial flutter | an average of 24 months following the ablation procedure
  Recurrence rate of typical atrial flutter
Rate of occurrence of atypical flutter | an average of 24 months following the ablation procedure
  Occurrence rate of atypical flutter defined as a continuous atrial activity (with no return to the isoelectric line)in at least one lead, whose ECG appearance of F waves is different from that of a typical flutter
Rate of occurrence of atrial tachycardia | an average of 24 months following the ablation procedure
  Rate of occurrence of atrial tachycardia defined as an atrial activaty that generates a P wave with return to the isoelectric line in all leads
Rate of complications related to the ablation procedure | an average of 3 months after the ablation procedure
  The following complications will be considered:
  Hematoma at punction site, Thromboembolic accident, Tamponnade, Phrenic nerve paralysis, Symptomatic stenosis of pulmonary vein, Atrio-ventricular block Atrioesophageal fistula
Rate of major cardiovascular events | an average of 24 months following the ablation procedure
  Rate of major cardiovascular events such as rehospitalization for arrhythmia, heart failure, or embolic accident
All mortality rate | an average of 24 months following the ablation procedure
  All mortality rate (including sudden death and any type of death)

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Anselme, MD, Principal Investigator — University Hospital, Rouen
Locations (15):
- France (15):
  - CHU de Brest, Brest
  - CHU Grenoble, Grenoble
  - CH La Rochelle, La Rochelle
  - AP-HM - Hôpital Nord, Marseille
  - Hôpital Privé de Clairval, Marseille
  - CHU de Nantes, Nantes
  - Nouvelles Cliniques Nantaises, Nantes
  - CHU de Rennes, Rennes
  - University Hospital of Rouen, Rouen
  - CHU de Strasbourg, Strasbourg
  - Clinique Pasteur, Toulouse
  - CHU de Tours, Tours
  - Clinique Saint Gatien, Tours
  - Clinique Saint Joseph, Trélazé
  - Polyclinique Vauban, Valenciennes